CLINICAL TRIAL: NCT03255876
Title: Effects of Enriched Fruit Juice on Blood Glucose Levels After a Meal in Healthy Subjects
Acronym: PolyGlucHeal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Gary Williamson, Professor Gary Williamson, University of Leeds
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MEEC 16-011
Record Dates: First submitted 2017-08-17; First posted 2017-08-21 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Hyperglycemia, Postprandial; Healthy
Keywords: Polyphenols; Hyperglycemia; Postprandial; Starch; Alpha-amylase
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enriched pomegranate juice (Experimental): Participants will consume 200 ml of pure pomegranate juice enriched with grape seed and apple peel extracts concomitantly with 109 g of white bread
  Interventions: Dietary Supplement: Enriched pomegranate juice
- Placebo beverage (Placebo Comparator): Participants will consume 200 ml of placebo drink concomitantly with 109 g of white bread
  Interventions: Dietary Supplement: Placebo beverage

INTERVENTIONS:
Dietary Supplement: Enriched pomegranate juice — Pure pomegranate juice enriched with grape seed and apple peel extract (200 ml) to be consumed with 109 g of bread
  Arms: Enriched pomegranate juice
Dietary Supplement: Placebo beverage — Beverage containing the same type and amount of carbohydrates as pomegranate juice and similar flavor (200 ml) to be consumed with 109 g of bread
  Arms: Placebo beverage

SUMMARY:
Results from a large number of studies in humans have shown that diets rich in foods that give lower glucose response bring lower risk of type 2 diabetes. Polyphenols, naturally found in fruits, vegetables and grains, have shown the potential to attenuate post-prandial blood glucose spikes following a carbohydrate-rich meal, through partial inhibition of the main enzymes of carbohydrate digestion and reduction in glucose and fructose transport from the gut after digestion and by enhancing the insulin action after glucose reaches the bloodstream.

This study is designed to determine whether polyphenols, as normally and naturally present in food extracts and beverages, added to a carbohydrate-rich meal, can lower blood glucose levels after its consumption, and hence lower its glycaemic index, and if this effect is mediated through effects on insulin and other hormones. The study is designed as an acute, double-blind, randomised, placebo-controlled crossover trial in 24 healthy subjects with normal glycaemic response to white bread. Participants will be asked to consume either white bread with pomegranate juice enriched with extracts from grape seeds and apple peels or white bread with placebo drink. The effects on plasma glucose levels, levels of hormones and other biomarkers involved in postprandial response will be determined over 3 hours after the consumption.

DETAILED DESCRIPTION:
Consumption of carbohydrate-rich foods or sugary drinks affects blood glucose levels. Results from a large number of studies in humans have shown that diets rich in foods that give lower glucose response beneficially affect elevated fasting blood glucose and insulin levels, increase the sensitivity to insulin, contribute to the reduction of body weight and lipids levels and ultimately bring lower risk of type 2 diabetes.

Blood glucose responses depend on the amount and type of carbohydrate(s) present in the meal. Difference in post-prandial blood glucose response to different types of carbohydrates is mainly due to the different rate of their digestion. However, response to the same carbohydrate-rich food can be different between different individuals. Blood glucose levels after carbohydrate-rich meal are shown to be significantly higher in subjects on high-fat diet, in overweight or obese people, or in subjects with different levels of digestive enzymes.

Results from in vitro studies indicate the potential of polyphenols, naturally found in fruits, vegetables and grains, to attenuate post-prandial blood glucose spikes following a carbohydrate-rich meal. It was previously shown that different polyphenols can slow down carbohydrate digestion through partial inhibition of the main enzymes involved, can decrease glucose and fructose transport from the gut after digestion and can improve the action of insulin after glucose reaches the bloodstream.

In the previous study it was shown that pomegranate juice attenuates the increase in blood glucose levels after a starchy meal. This effect is, at least partly, the result of hindered starch digestion by polyphenols present in pomegranate juice.

The present study will determine whether polyphenols, as normally and naturally present in food extracts and beverages, added to a carbohydrate-rich meal, can lower blood glucose levels after its consumption, and hence lower its glycaemic index, and if this effect is mediated through effects on insulin and other hormones or determined by the individual levels of digestive enzymes.

Healthy volunteers will be asked to consume two different meals: (1) white bread with pomegranate juice enriched with extracts from grape seeds and apple peels or (2) white bread with placebo drink with the same type and amount of carbohydrates and similar flavor as enriched pomegranate juice, but without polyphenols.

The levels of glucose, insulin, gastric inhibitory polypeptide (GIP) and glucagon like peptide-1 (GLP-1) will be measured in plasma isolated from blood samples obtained before and up to 3 hours after the consumption of each meal. The levels of triglycerides and relevant organic and fatty acids will also be determined.

Before recruitment volunteers will be screened for eligibility based on glucose levels, BMI and glycemic response to white bread. Additional measurements taken at the screening will include blood pressure values and blood lipids levels. All participants will be characterized for the activity of salivary a-amylase and copies of a-amylase gene (AMY1).

ELIGIBILITY:
Inclusion Criteria:

* Fasting glucose ≤ 5.6 mM;
* Body mass index (BMI) ≤ 30;
* Max glucose after the consumption of app. 109g of white bread less than about 8-9 mM (which is typical for the subjects we have measured previously);

Exclusion Criteria:

* Smoking;
* Participating in another trial that requires blood collection;
* Diagnosed with any chronic illness (including diabetes, hypertension etc.);
* On long term prescribed medication (except contraceptives);
* Pregnant or lactating;
* On a special diet or dietary regimen (for weight management or if regularly consuming fruit extract supplements);
* Allergy to fruits vegetables or pollen.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-04-10 (Actual); Primary Completion 2018-08-20 (Estimated); Study Completion 2018-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes in maximal incremental plasma glucose level (iCmax) between baseline and endpoint within the intervention group vs. placebo control. | Baseline, 15 min, 30 min, 45 min, 60 min, 90 min, 120 min, 150 min, 180 min.
  The incremental glucose levels will be determined for each time point (at 15, 30, 45, 60, 90, 120, 150 and 180 min) as the change in plasma glucose levels after the consumption of enriched pomegranate juice or placebo drink concomitantly with white bread, compared to the glucose levels before the consumption of test meals (baseline value, t=0min).

SECONDARY OUTCOMES:
Changes in area under the curve of incremental plasma glucose levels (iAUC) in the intervention group vs. placebo control. | Baseline, 15 min, 30 min, 45 min, 60 min, 90 min, 120 min, 150 min, 180 min.
  The glucose iAUC will be determined from all incremental plasma glucose levels at the defined time points (0, 15, 30, 45, 60, 90, 120, 150 and 180 min) after the consumption of test and control meals based on trapezoid rule.
Changes in plasma insulin levels between baseline and endpoint within the intervention group vs. placebo control. | Baseline, 15 min, 30 min, 45 min, 60 min, 90 min, 120 min, 150 min, 180 min.
  Insulin levels measured at the baseline and at each time point (at 15, 30, 45, 60, 90,120, 150 and 180 min) after the consumption of test and control meals.
Changes in plasma gastric inhibitory peptide (GIP) levels between baseline and endpoint within the intervention group vs. placebo control. | Baseline, 15 min, 30 min, 45 min, 60 min, 90 min, 120 min, 150 min, 180 min.
  GIP levels measured in plasma at the baseline and at each time point (at 15, 30, 45, 60, 90,120, 150 and 180 min) after the consumption of test and control meals.
Changes in glucagon-like peptide-1 (GIP-1) levels between baseline and endpoint within the intervention group vs. placebo control. | Baseline, 15 min, 30 min, 45 min, 60 min, 90 min, 120 min, 150 min, 180 min.
  GLP-1 levels measured in plasma at the baseline and at each time point (at 15, 30, 45, 60, 90,120, 150 and 180 min) after the consumption of test and control meals.

OTHER OUTCOMES:
Changes in organic acids profile between baseline and endpoint within the intervention group vs. placebo control. | Baseline, 15 min, 30 min, 45 min, 60 min, 90 min, 120 min, 150 min, 180 min.
  Levels of selected organic acids measured in plasma at the baseline and at each time point (at 15, 30, 45, 60, 90,120, 150 and 180 min) after the consumption of test and control meals.
Changes in fatty acids profile between baseline and endpoint within the intervention group vs. placebo control. | Baseline, 15 min, 30 min, 45 min, 60 min, 90 min, 120 min, 150 min, 180 min.
  Levels of selected free-fatty acids measured in serum at the baseline and at each time point (at 15, 30, 45, 60, 90,120, 150 and 180 min) after the consumption of test and control meals.
Changes in triglycerides levels between baseline and endpoint within the intervention group vs. placebo control. | Baseline, 15 min, 30 min, 45 min, 60 min, 90 min, 120 min, 150 min, 180 min.
  Levels of triglycerides measured in serum at the baseline and at each time point (at 15, 30, 45, 60, 90,120, 150 and 180 min) after the consumption of test and control meals.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Williamson, PhD, Study Chair — University of Leeds; Aleksandra Konic Ristic, PhD, Principal Investigator — University of Leeds
Locations (1):
- School of Food Science and Nutrition, University of Leeds, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes